CLINICAL TRIAL: NCT04789512
Title: Evaluation of Respiratory Muscle Strength and Pulmonary Functions in Volleyball Players Suffering From Covid-19
Brief Title: Respiratory Muscle Strength in Volleyball Players Suffered From COVID-19
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Zeliha ÇELİK, Research assistant, Gazi University
Other Study IDs: 2021-189
Record Dates: First submitted 2021-03-06; First posted 2021-03-09 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: respiratory muscles; pulmonary functions
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid-19 players: Female volleyball players with Covid-19
  Interventions: Other: Respiratory functions
- non-Covid-19 players: Female volleyball players with non Covid-19
  Interventions: Other: Respiratory functions

INTERVENTIONS:
Other: Respiratory functions — Respiratory muscle strength, pulmonary functions and body composition were evaluated in volleyball players

SUMMARY:
In literature, there is no data evaluating respiratory functions in volleyball players during Covid-19 pandemic. The aim of this study is to evaluate and compared pulmonary functions, respiratory muscle strength, body compositions and performance situations perceptions in female volleyball players with Covid-19 and non-Covid-19.

ELIGIBILITY:
Inclusion Criteria:

* having passed at least 30 days after the Polymerase Chain Reaction (PCR) test turned negative
* willing to participate in the study

Exclusion Criteria:

* having a history of chronic lung disease
* unwilling to participate in the study

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Female volleyball players
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle strength | 10 minute
  Maximal inspiratory and expiratory muscle strength will be evaluated using mouth pressure device.

SECONDARY OUTCOMES:
FEV1 | 5 minute
  Pulmonary function tests will be performed using a spirometry according to the American Thoracic Society and European Respiratory Society criteria. FEV1 will be evaluated. The percentage of predicted value <70% will be expressed as abnormal.
FVC | 5 minute
  Pulmonary function tests will be performed using a spirometry according to the American Thoracic Society and European Respiratory Society criteria. FVC will be evaluated. The percentage of predicted value <70% will be expressed as abnormal
FEV1/FVC | 5 minute
  Pulmonary function tests will be performed using a spirometry according to the American Thoracic Society and European Respiratory Society criteria. FEV1/FVC will be evaluated.
PEF | 5 minute
  Pulmonary function tests will be performed using a spirometry according to the American Thoracic Society and European Respiratory Society criteria. PEF will be evaluated. The percentage of predicted value <70% will be expressed as abnormal.
FEF2575 | 5 minute
  Pulmonary function tests will be performed using a spirometry according to the American Thoracic Society and European Respiratory Society criteria. FEF2575 will be evaluated. The percentage of predicted value <50% will be expressed as abnormal.
Fat mass | 2 minute
  Fat mass will be evaluated using TANITA bioelectrical impedance analysis.
Fat mass percent | 2 minute
  Fat mass percent will be evaluated using TANITA bioelectrical impedance analysis.
Fat-free mass | 2 minute
  Fat-free mass will be evaluated using TANITA bioelectrical impedance analysis.
Body mass index | 2 minute
  Body mass index will be evaluated using TANITA bioelectrical impedance analysis.
Predicted muscle mass | 2 minute
  Predicted muscle mass will be evaluated using TANITA bioelectrical impedance analysis.
Symptom severity perceptions | 1 minute
  Symptom severity perceptions will be evaluated Numeric Rating Scale.The severity of symptoms perceptions related to Covid are scored 0-10 point. Higher scores indicate higher severity of symptoms.
Performance situations perceptions | 1 minute
  Performance situations perceptions will be evaluated Numeric Rating Scale. Performance situations perceptions of all players are also scored 0-10 point. Higher scores indicate greater performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Celik Z, Guzel NA, Kafa N, Kokturk N. Respiratory muscle strength in volleyball players suffered from COVID-19. Ir J Med Sci. 2022 Oct;191(5):1959-1965. doi: 10.1007/s11845-021-02849-z. Epub 2021 Nov 8. PMID 34748144